CLINICAL TRIAL: NCT01840254
Title: Effect of Combination Dexmedetomidine Added to Fentanyl-based Intravenous Patient-controlled Analgesia on Nausea Vomiting in Highly Susceptible Patients Undergoing Lumbar Spinal Surgery: Prospective Double Blinded Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0490
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: PONV
Keywords: PONV; IV PCA; dexmedetomidine; Female; non-smoking; lumbar spine surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): addition of dexmedetomidine to fentanyl-based intravenous patient controlled analgesia (PCA)
  Interventions: Drug: dexmedetomidine
- normal saline (Placebo Comparator): normal saline as a placebo
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: dexmedetomidine
  Arms: dexmedetomidine
Drug: normal saline
  Arms: normal saline

SUMMARY:
The aim of this study is to test the hypothesis that addition of dexmedetomidine to fentanyl-based intravenous patient controlled analgesia (PCA) reduces requirement of fentanyl bolus and consequent postoperative nausea and vomiting in high-risk patients undergoing lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

1. female, non-smoking patient who are 20-65 of age scheduled for elective lumbar spine surgery

Exclusion Criteria:

1. Bradycardia on EKG (45bpm)
2. Atrioventricular conduction disorder
3. Uncontrolled hypertension
4. angina history
5. obesity (BMI ≥ 30 kg/m2)
6. Preoperative administration of opioid
7. Preoperative administration of antiemetics
8. Gastrointestinal disorder history
9. Hepatic or renal disease
10. Pregnant 11. Foreigner

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
total dose and bolus administration of opioid | an expected average of 48 hrs for requirements of total dose and number of bolus administration of PCA
  After induction of anesthesia, peak velocity of carotid artery blood flow is measured by the pulsed wave Doppler signal obtained from the left common carotid artery. Respirophasic variation of the peak velocity is defined as the difference between the maximum and the minimum values of peak velocity divided by the mean of the two values during one respiratory cycle. Fluid responder is defined as a patient whose stroke volume index is increased ≥15% after volume expansion. The receiver operating characteristic curve analysis to discriminiate fludi responder is performed.

SECONDARY OUTCOMES:
consequent postoperative nausea and vomiting | an expected average of 48 hrs for assessing of the 11-points verbal numerical rating scales
  After induction of anesthesia, peak velocity of carotid artery blood flow is measured by the pulsed wave Doppler signal obtained from the left common carotid artery. Respirophasic variation of the peak velocity is defined as the difference between the maximum and the minimum values of peak velocity divided by the mean of the two values during one respiratory cycle. Fluid responder is defined as a patient whose stroke volume index is increased ≥15% after volume expansion. The receiver operating characteristic curve analysis to discriminate fluid responder is performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Song Y, Shim JK, Song JW, Kim EK, Kwak YL. Dexmedetomidine added to an opioid-based analgesic regimen for the prevention of postoperative nausea and vomiting in highly susceptible patients: A randomised controlled trial. Eur J Anaesthesiol. 2016 Feb;33(2):75-83. doi: 10.1097/EJA.0000000000000327. PMID 26258655